CLINICAL TRIAL: NCT04894656
Title: Assessing Intestinal Barrier Function and Permeability in Patients With Gastroparesis
Brief Title: Intestinal Permeability and Gastroparesis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn due to funding.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David J. Cangemi, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-000771
Record Dates: First submitted 2021-05-11; First posted 2021-05-20 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Gastroparesis; Healthy
MeSH Terms: conditions — Gastroparesis | interventions — Urinalysis; Gastroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastroparesis patients (Experimental)
  Interventions: Diagnostic Test: Labs, urine tests, upper endoscopy with biopsy and confocal laser endomicroscopy
- Healthy volunteers (Active Comparator)
  Interventions: Diagnostic Test: Labs, urine tests, upper endoscopy with biopsy and confocal laser endomicroscopy

INTERVENTIONS:
Diagnostic Test: Labs, urine tests, upper endoscopy with biopsy and confocal laser endomicroscopy — Tests to assess intestinal permeability

SUMMARY:
The purpose of this study is to investigate potential mechanisms that could lead to the development of a condition known as gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-75 years old).
* Men and women.
* Patients with gastroparesis.

Exclusion Criteria:

* Patients will be excluded from the study if symptoms are thought to represent an organic disorder (e.g., peptic ulcer disease, hepatitis, pancreatitis, inflammatory bowel disease, a known malignancy, radiation-induced injury, an active infection, vasculitis, celiac disease), GERD, esophagitis, eosinophilic esophagitis or H. pylori.
* Patients with uncontrolled diabetes mellitus (hemoglobin A1C > 10).
* Patients with prior surgery to the esophagus, stomach or duodenum.
* Patients taking opioids, steroids, anti-histamines, immunosuppressive agents, NSAIDs, or mast cell stabilizing agents within the prior 3 months.
* Patients currently prescribed aspirin or aspirin regimens for other clinical reasons.
* Patients with known allergies to lactulose: mannitol will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Assess duodenal epithelial tight junction structure in GP patients using confocal laser endomicroscopy. | through study completion, approximately 3-4 days

SECONDARY OUTCOMES:
Assess small intestinal permeability using the lactulose:mannitol urinary excretion test. | through study completion, approximately 3-4 days
Measure serum levels of immune markers (e.g., IL-1,4,6,10,12,13,18; zonulin, CRP, TNF-alpha, tryptase,) in GP patients and compare to healthy controls. | One time measurement
Quantitate different duodenal cell types (e.g., mast cells (CK117), eosinophils, enterochromaffin, intraepithelial lymphocytes (IELs) and CCK-containing cells) in patients with GP using biopsies from both the D1 and D2 duodenal segments. | through study completion, approximately 3-4 days
Assess the relationship of GP symptoms to intestinal permeability, using validated questionnaires, and to histopathological changes. | through study completion, approximately 3-4 days

CONTACTS AND LOCATIONS:
Overall Officials: David Cangemi, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials